CLINICAL TRIAL: NCT01418235
Title: A Phase 1 Placebo-controlled Clinical Trial to Evaluate the Safety and Immunogenicity of SAAVI DNA-C2, SAAVI MVA-C and Novartis Subtype C gp140 With MF59 Adjuvant in Various Vaccination Schedules in HIV-uninfected Healthy Vaccinia-naïve Adult Participants in South Africa
Brief Title: Safety of and Immune Response to a DNA HIV Vaccine Boosted With a Modified Vaccinia HIV Vaccine and Protein HIV Vaccine in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: HIV Vaccine Trials Network (Network)
Collaborators: South Africa AIDS Vaccine Initiative (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: HVTN 086/SAAVI 103
Record Dates: First submitted 2011-06-17; First posted 2011-08-17 (Estimated); Last update posted 2019-06-21 (Actual); Status verified 2019-06

CONDITIONS: HIV Seronegativity; HIV Preventive Vaccine
Keywords: HIV Infections; Acquired Immunodeficiency Syndrome; Lentivirus Infections; Retroviridae Infections; RNA Virus Infections; Virus Diseases; Sexually Transmitted Diseases, Viral; Sexually Transmitted Diseases; Immunologic Deficiency Syndromes; Immune System Diseases; Slow Virus Diseases
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome; Lentivirus Infections; Retroviridae Infections; RNA Virus Infections; Virus Diseases; Sexually Transmitted Diseases, Viral; Sexually Transmitted Diseases; Immunologic Deficiency Syndromes; Immune System Diseases; Slow Virus Diseases

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Group 1: MVA-C + gp140/MF59 (Experimental)
  Interventions: Biological: MVA-C + gp140/MF59
- Group 2: MVA-C + gp140/MF59 (Experimental)
  Interventions: Biological: MVA-C + gp140/MF59
- Group 3: DNA-C2 + MVA-C (Experimental)
  Interventions: Biological: DNA-C2 + MVA-C
- Group 4: DNA-C2 + MVA-C + gp140/MF59 (Experimental)
  Interventions: Biological: DNA-C2 + MVA-C + gp140/MF59

INTERVENTIONS:
Biological: MVA-C + gp140/MF59 — SAAVI MVA-C administered as 0.5 ml intramuscularly in right deltoid, with placebo in left deltoid, at Month 0; SAAVI MVA-C administered as 0.5 ml intramuscularly in right deltoid at Month 1; Novartis subtype C gp140 admixed with Novartis MF59 adjuvant administered as 0.5 ml intramuscularly in left deltoid, with placebo in right deltoid, at Months 3, 6.
  Placebo comparator: Placebo administered at Months 0, 1, 3, 6
  Arms: Group 1: MVA-C + gp140/MF59
Biological: MVA-C + gp140/MF59 — SAAVI MVA-C administered as 0.5 ml intramuscularly in right deltoid, with Novartis subtype C gp140 admixed with Novartis MF59 adjuvant administered as 0.5 ml intramuscularly in left deltoid, at Months 0, 3; placebo in right deltoid at Month 1; placebo in each deltoid at Month 6
  Placebo comparator: Placebo administered at Months 0, 1, 3, 6
  Arms: Group 2: MVA-C + gp140/MF59
Biological: DNA-C2 + MVA-C — SAAVI DNA-C2 administered as 1 ml intramuscularly in right deltoid, with placebo in left deltoid, at Month 0; SAAVI DNA-C2 administered as 1 ml intramuscularly in right deltoid at Month 1; SAAVI MVA-C administered as 0.5 ml intramuscularly in right deltoid, with placebo in left deltoid, at Months 3, 6
  Placebo comparator: Placebo administered at Months 0, 1, 3, 6
  Arms: Group 3: DNA-C2 + MVA-C
Biological: DNA-C2 + MVA-C + gp140/MF59 — SAAVI DNA-C2 administered as 1 ml intramuscularly in right deltoid, with placebo in left deltoid, at Month 0; SAAVI DNA-C2 administered as 1 ml intramuscularly in right deltoid at Month 1; SAAVI MVA-C administered as 0.5 ml intramuscularly in right deltoid at Months 3, 6; Novartis subtype C gp140 admixed with Novartis MF59 adjuvant administered as 0.5 ml intramuscularly in left deltoid, with placebo in right deltoid, at Months 3, 6
  Placebo comparator: Placebo administered at Months 0, 1, 3, 6
  Arms: Group 4: DNA-C2 + MVA-C + gp140/MF59

SUMMARY:
Sub-Saharan Africa is the region most affected by the global Human Immunodeficiency Virus (HIV) epidemic. A vaccine is the most promising preventive approach against new HIV infections. The purpose of this study is to evaluate the safety and immunogenicity of 4 experimental preventive HIV vaccine regimens in HIV-uninfected adults in South Africa.

DETAILED DESCRIPTION:
The worldwide Human Immunodeficiency Virus / Acquired Immunodeficiency Syndrome (HIV/AIDS) epidemic may only be controlled through development and utilization of a safe and effective vaccine that will prevent HIV infection. Due to the high prevalence of HIV-1 subtype C in southern Africa, the South African AIDS Vaccine Initiative (SAAVI), the HIV Vaccine Trials Network (HVTN), Novartis, and the National Institute of Allergy and Infectious Diseases (NIAID) are evaluating three subtype C HIV vaccines, SAAVI DNA-C2, SAAVI MVA-C, and Novartis Subtype C gp140 through this study. These vaccines will be used together in four prime-boost regimens. The SAAVI DNA-C2 vaccine is a multigene deoxyribonucleic acid (DNA) vaccine consisting of two DNA plasmids in equal amounts that express an HIV-1 subtype C polyprotein comprising of Gag-Reverse Transcriptase-Tat-Nef and an HIV-1 subtype C truncated Env. SAAVI MVA-C is a recombinant modified vaccinia Ankara (MVA) vaccine expressing the same immunogens as the SAAVI DNA-C2 vaccine. MVA is a highly attenuated vaccinia virus. The Novartis protein subunit vaccine is a Subtype C oligomeric V2 loop deleted glycoprotein 140 (gp140) vaccine (gp140[delta]V2.TV1), given with MF59 adjuvant.

This trial is designed to build upon the Thai RV144 HIV vaccine trial, which demonstrated an efficacy of 31.2% among participants who received a different vaccine regimen of a pox prime followed by a concurrently-administered protein boost. This primary purpose of HVTN 086 is to evaluate the safety and immunogenicity of SAAVI DNA-C2, SAAVI MVA-C and Novartis Clade C gp140TV1ΔV2 with MF59 adjuvant in various vaccination regimens. The primary analysis will focus on a ranking strategy of the vaccine regimens that is guided by measurements of the immune responses elicited by these vaccines and their respective modes of delivery in various combinations, both sequential and concurrent.

Participants will actively participate in this study for 12 months. Participants will be randomly assigned to receive either a prime-boost preventive vaccine regimen or placebo. Four prime-boost preventive vaccine regimens will be compared; each participant will be randomized to one of 4 groups. Participants in Group 1 will receive MVA-C at months 0 and 1, and gp140/MF59 at months 3 and 6. Group 2 will receive MVA-C and gp140/MF59 at months 1 and 3. Group 3 will receive DNA-C at months 0 and 1, and MVA-C at months 3 and 6. Group 4 will receive DNA-C at months 0 and 1, and both MVA-C and gp140/MF59 at months 3 and 6. Additional study visits will occur at Weeks 2, 6, 13, 14, 26, 28, 36, and 48. All participants will be contacted once annually for 3 years and asked questions about their health. Study procedures include physical exams, blood and urine collection, HIV testing, an electrocardiogram, and questionnaire. Some blood collected from participants will be stored and used in future research. Risk-reduction counseling will be conducted at all study visits.

ELIGIBILITY:
Inclusion Criteria:

1. Age of 18 to 45 years
2. Access to a participating HVTN clinical research site and willingness to be followed for the planned duration of the study
3. Ability and willingness to provide informed consent
4. Assessment of understanding: volunteer demonstrates understanding of this study and other relevant study results and completes a questionnaire prior to first vaccination with verbal demonstration of understanding of all questionnaire items answered incorrectly
5. Willingness to receive HIV test results
6. Willingness to discuss HIV infection risks, amenable to HIV risk reduction counseling, and committed to maintaining behavior consistent with low risk of HIV exposure through the last required protocol clinic visit
7. Assessed by clinic staff as being at "low risk" for HIV infection on the basis of sexual behavior within the 12 months prior to enrollment defined as follows:

   * Sexually abstinent, or
   * In a mutually monogamous relationship with a partner with a known HIV-uninfected status, or
   * Had one partner believed to be HIV-uninfected with whom he/she regularly used condoms for vaginal and anal intercourse
8. Willing to be contacted annually after completion of scheduled clinic visits for a total of 3 years following initial study injection
9. Agrees not to enroll in another study of an investigational research agent prior to completion of last required protocol clinic visit (excludes annual contacts for safety surveillance)
10. Good general health as shown by medical history, physical exam, and screening laboratory tests
11. Hemoglobin = 11.0 g/dL for volunteers who were born female, = 13.0 g/dL for volunteers who were born male
12. White blood cell (WBC) count = 3,300 to 12,000 cells/mm3
13. Total lymphocyte count = 800 cells/mm3
14. Platelets = 125,000 to 550,000/mm3
15. Chemistry panel: Alanine aminotransferase (ALT), aspartate aminotransferase (AST), and alkaline phosphatase < 1.25 times the institutional upper limit of normal
16. Cardiac Troponin T (cTnT) does not exceed the institutional upper limit of normal
17. Negative HIV-1 and -2 blood test: Sites may use locally available assays that have been approved by HVTN Laboratory Operations.
18. Negative Hepatitis B surface antigen (HBsAg)
19. Negative anti-Hepatitis C virus antibodies (anti-HCV), or negative HCV polymerase chain reaction (PCR) if the anti-HCV is positive
20. Normal urine:

    * Negative urine glucose, and
    * Negative or trace urine protein, and
    * Negative or trace urine hemoglobin (if trace hemoglobin is present on dipstick, a microscopic urinalysis within institutional normal range).
21. Volunteers who were born female: negative serum or urine beta human chorionic gonadotropin (ß-HCG) pregnancy test performed prior to vaccination on the day of initial vaccination
22. Reproductive status: A volunteer who was born female must:

    * Agree to consistently use effective contraception, from at least 21 days prior to enrollment through 90 days after the participant's last vaccination, for sexual activity that could lead to pregnancy. Effective contraception for participants in South Africa is defined as using 2 methods, including 1 of the following:
    * Condoms (male or female) with or without a spermicide,
    * Diaphragm or cervical cap with spermicide,

    PLUS 1 of the following methods:
    * Intrauterine device (IUD),
    * Hormonal contraception, or
    * Successful vasectomy in the male partner (considered successful if a volunteer reports that a male partner has [1] documentation of azoospermia by microscopy, or [2] a vasectomy more than 2 years ago with no resultant pregnancy despite sexual activity postvasectomy);
    * Or not be of reproductive potential, such as having reached menopause (no menses for 1 year) or having undergone hysterectomy, bilateral oophorectomy, or tubal ligation;
    * Or be sexually abstinent.
23. Volunteers who were born female must also agree not to seek pregnancy through alternative methods, such as artificial insemination or in vitro fertilization until after the last required protocol clinic visit

Exclusion Criteria:

1. Vaccinia (smallpox) vaccination determined by: (1) clinical evidence of vaccinia scarification; (2) self-reported history of vaccinia vaccination; or (3) birth year 1977 or earlier. (Not excluded: a participant born in or before 1977 who self reports he/she did not receive vaccinia [smallpox] vaccination and has no evidence of scarification.)
2. Within the 12 months prior to enrollment: excessive daily alcohol use or frequent binge drinking or chronic marijuana abuse or any other use of illicit drugs
3. Within the 12 months prior to enrollment: a history of newly acquired syphilis, gonorrhea, non-gonococcal urethritis, herpes simplex virus type 2 (HSV2), Chlamydia, pelvic inflammatory disease (PID), trichomonas, mucopurulent cervicitis, epididymitis, proctitis, lymphogranuloma venereum, chancroid, or hepatitis B
4. Untreated or incompletely treated syphilis infection
5. HIV vaccine(s) received in a prior HIV vaccine trial. For potential participants who have received control/placebo in an HIV vaccine trial, the HVTN 086 / SAAVI 103 PSRT will determine eligibility on a case-by-case basis.
6. Non-HIV experimental vaccine(s) received within the last 5 years in a prior vaccine trial. Exceptions may be made for vaccines that have subsequently undergone licensure by the FDA or MCC. For potential participants who have received control/placebo in an experimental vaccine trial, the HVTN 086 / SAAVI 103 PSRT will determine eligibility on a case-by-case basis. For potential participants who have received an experimental vaccine(s) greater than 5 years ago, eligibility for enrollment will be determined by the PSRT on a case-by-case basis.
7. Immunosuppressive medications received within 168 days before first vaccination. (Not excluded: [1] corticosteroid nasal spray for allergic rhinitis; [2] topical corticosteroids for mild, uncomplicated dermatitis; or [3] oral/parenteral corticosteroids given for non-chronic conditions not expected to recur [length of therapy 10 days or less with completion at least 30 days prior to enrollment].)
8. Blood products received within 120 days before first vaccination
9. Immunoglobulin received within 60 days before first vaccination
10. Live attenuated vaccines (not including influenza vaccine) received within 30 days before first vaccination or scheduled within 14 days after injection (eg, measles, mumps, and rubella [MMR]; oral polio vaccine [OPV]; varicella; yellow fever)
11. Influenza vaccine or any vaccines that are not live attenuated vaccines and were received within 14 days prior to first vaccination (eg, tetanus, pneumococcal, Hepatitis A or B)
12. Investigational research agents received within 30 days before first vaccination or scheduled within 14 days after vaccination
13. Allergy treatment with antigen injections within 30 days before first vaccination or that are scheduled within 14 days after first vaccination
14. Current anti-tuberculosis (TB) prophylaxis or therapy
15. Clinically significant medical condition, physical examination findings, clinically significant abnormal laboratory results, or past medical history with clinically significant implications for current health. A clinically significant condition or process includes but is not limited to:

    * A process that would affect the immune response,
    * A process that would require medication that affects the immune response,
    * Any contraindication to repeated injections or blood draws,
    * A condition that requires active medical intervention or monitoring to avert grave danger to the participant's health or well-being during the study period,
    * A condition or process for which signs or symptoms could be confused with reactions to vaccine, or
    * Any condition specifically listed among the exclusion criteria below.
16. Any medical, psychiatric, occupational, or other condition that, in the judgment of the investigator, would interfere with, or serve as a contraindication to, protocol adherence, assessment of safety or reactogenicity, or a participant's ability to give informed consent.
17. Serious adverse reactions to vaccines including anaphylaxis and related symptoms such as hives, respiratory difficulty, angioedema, and/or abdominal pain. (Not excluded: a participant who had a nonanaphylactic adverse reaction to pertussis vaccine as a child.)
18. Hypersensitivity to eggs or egg products
19. ECG with clinically significant findings, or features that would interfere with the assessment of myo/pericarditis, as determined by a contract ECG laboratory or cardiologist, including any of the following: (1) conduction disturbance (complete left or complete right bundle branch block or nonspecific intraventricular conduction disturbance with QRS =120ms, AV block of any degree, or QTc prolongation (> 440ms); (2) repolarization (ST segment or T wave) abnormality; (3) significant atrial or ventricular arrhythmia; (4) frequent atrial or ventricular ectopy (eg, frequent premature atrial contractions, 2 premature ventricular contractions in a row); (5) ST elevation consistent with ischemia; (6) evidence of past or evolving myocardial infarction.
20. Cardiac risk factors, including 2 or more of the following: (1) participant report of history of elevated blood cholesterol defined as fasting low density lipoprotein (LDL) > 160 mg/dL; (2) first degree relative (eg, mother, father, brother, or sister) who had coronary artery disease before the age of 50 years; (3) current smoker; or (4) BMI = 35.
21. History of, or known active cardiac disease including: (1) previous myocardial infarction (heart attack); (2) angina pectoris; (3) congestive heart failure; (4) valvular heart disease including mitral valve prolapse; (5) cardiomyopathy; (6) pericarditis; (7) stroke or transient ischemic attack; (8) chest pain or shortness of breath with activity (such as walking up stairs); (9) dysrhythmia/episodic palpitations (Not excluded: sinus arrhythmia); or (10) other heart conditions under the care of a doctor.
22. Autoimmune disease
23. Immunodeficiency
24. Asthma other than mild, well-controlled asthma. Exclude a participant who:

    * Generally uses a bronchodilator (beta2 agonist) daily, or
    * In the past year, has (any of the following):
    * Had > 1 exacerbation of symptoms treated with oral steroids (Note: oral/parenteral steroid use for asthma is exclusionary within 168 days before first vaccination.);
    * Routinely used moderate to high dose inhaled corticosteroids (eg, more than the equivalent of 250 µg fluticasone; 400 µg budesonide; 500 µg beclomethasone; or 1000 µg triamcinolone/flunisolide, as a daily dose) or theophylline for asthma; or
    * Needed emergency care, urgent care, hospitalization, or intubation for asthma.
25. Diabetes mellitus type 1 or type 2, including cases controlled with diet alone. (Not excluded: history of isolated gestational diabetes.)
26. Thyroidectomy, or thyroid disease requiring medication during the last 12 months
27. Angioedema within the last 3 years if episodes are considered serious or have required medication within the last 2 years
28. Hypertension:

    * If a person has been diagnosed with hypertension during screening or previously, exclude for hypertension that is not well controlled. Well-controlled hypertension is defined as blood pressure consistently = 140 mm Hg systolic and = 90 mm Hg diastolic, with or without medication, with only isolated, brief instances of higher readings, which must be = 150 mm Hg systolic and = 100 mm Hg diastolic. For these participants, blood pressure must be = 140 mm Hg systolic and = 90 mm Hg diastolic at enrollment.
    * If a person has NOT been diagnosed with hypertension during screening or previously, exclude for systolic blood pressure = 150 mm Hg at enrollment or diastolic blood pressure = 100 mm Hg at enrollment.
29. Body mass index (BMI) = 40
30. Bleeding disorder diagnosed by a doctor (eg, factor deficiency, coagulopathy, or platelet disorder requiring special precautions)
31. Malignancy (Not excluded: a participant with a surgical excision and subsequent observation period that in the investigator's estimation has a reasonable assurance of sustained cure or is unlikely to recur during the period of the study.)
32. Seizure disorder (Not excluded: a participant with a history of seizures who has not required medications or had a seizure within the past 3 years.)
33. Asplenia: any condition resulting in the absence of a functional spleen
34. Psychiatric condition that precludes compliance with the protocol. Specifically excluded are persons with psychoses within the past 3 years, ongoing risk for suicide, or history of suicide attempt or gesture within the past 3 years.
35. Pregnant or breastfeeding

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 184 (Actual)
Dates: Start 2011-12-19 (Actual); Primary Completion 2013-10-07 (Actual); Study Completion 2015-12-09 (Actual)

PRIMARY OUTCOMES:
Signs and symptoms of local and systemic reactogenicity, laboratory measures of safety, and adverse events | Measured through approximately Month 12
Neutralizing antibody titers to tier 1 and tier 2 virus isolates as assessed by magnitude-breadth curves | Measured through approximately Month 12

SECONDARY OUTCOMES:
T-cell response rate and magnitude as detected by HIV-1 specific interferon-gamma/interleukin-2 intracellular cytokine staining | Measured 2 weeks after the 3rd and 4th vaccinations in Arms 1, 3, 4; measured 14 weeks after 2nd vaccination in Arm 2
Total HIV-1 Env-specific immunoglobulin G (IgG)-binding antibodies as determined by HIV-1 multiplex Ab assay ConS gp140, Du151 Env, and/or TV1gp140 specific IgG subclass (IgG1- IgG4) and IgA characterization determined by HIV-1 multiplex antibody assay | Measured 2 weeks after the 3rd and 4th vaccinations in Arms 1, 3, 4; measured 14 weeks after 2nd vaccination in Arm 2

CONTACTS AND LOCATIONS:
Overall Officials: Gavin Churchyard, Study Chair — Aurum Institute for Health Research
Locations (3):
- South Africa (3):
  - Perinatal HIV Research Unit, Johannesburg, Gauteng
  - Aurum Institute for Health Research, Klerksdorp, North West
  - Desmond Tutu HIV Centre, Cape Town, Western Cape

REFERENCES:
- [Derived] Churchyard G, Mlisana K, Karuna S, Williamson AL, Williamson C, Morris L, Tomaras GD, De Rosa SC, Gilbert PB, Gu N, Yu C, Mkhize NN, Hermanus T, Allen M, Pensiero M, Barnett SW, Gray G, Bekker LG, Montefiori DC, Kublin J, Corey L. Sequential Immunization with gp140 Boosts Immune Responses Primed by Modified Vaccinia Ankara or DNA in HIV-Uninfected South African Participants. PLoS One. 2016 Sep 1;11(9):e0161753. doi: 10.1371/journal.pone.0161753. eCollection 2016. PMID 27583368